CLINICAL TRIAL: NCT06422676
Title: Open-label Single-arm, Non-interventional, Multi-centre, Cohort Study for Evaluation of Clinical and Patient Reported Outcomes in New Users of BREZTRI (Budesonide / Glycopyrronium / Formoterol) in Routine Care Settings
Brief Title: MultIceNtre Non-intERVentional Study for Efficacy,Safety Evaluation of BREZTRI in Pts With COPD in RussiA
Acronym: MINERVA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00097
Record Dates: First submitted 2024-02-29; First posted 2024-05-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; COPD; BREZTRI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective-prospective, non-interventional, multi-centre study that will be conducted in routine clinical settings in Russia. Eligible patients with moderate to severe COPD routinely treated with BREZTRI will be observed according to routine clinical practice for up to 24 weeks.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a disease characterized by persistent airflow limitation that is usually progresses and is a consequence of a chronic inflammatory response of the respiratory pathways and lung tissue to the effects of inhaled harmful particles or gases. Exacerbations and comorbid conditions are an integral part of the disease and contribute significantly to the clinical picture and prognosis [1].

Patient-reported outcomes (both symptom-based and health-related quality of life-specific) are essential to evaluate symptoms, impact of symptoms on activities of daily living, and treatment response in COPD patients [12].

There is a need to evaluate the patient-reported outcomes during a triple therapy with budesonide + glycopyrronium bromide + formoterol (Breztri) in a real-life clinical practice. The aim of the study is to evaluate clinical and patient-reported outcomes of treatment with BREZTRI through effectiveness measures assessed pre- and post-treatment initiation and safety monitoring. The study results will be interpreted in the context of an open label, single arm study design where multiple factors, in addition to the new treatment, may contribute to the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-diagnosed COPD no less than 12 months before BREZTRI treatment start;
2. Patients who have not achieved adequate disease control when treated with a combination of ICS and LABA or a combination of LABA and LAMA
3. Initiated treatment with BREZTRI ≤12 weeks before inclusion as prescribed according to the label;
4. CAT score not more than 1 week before BREZTRI start is available;
5. Patients must be able and willing to read, comprehend and follow written instructions, and to comprehend and complete the questionnaires required by the protocol
6. Have signed a written Informed Consent Form (ICF).

Exclusion Criteria:

1. Documented COPD due to α-1 antitrypsin deficiency;
2. Previous treatment with triple fixed-dose combination in 12 months prior to inclusion;
3. Pregnancy or lactation period;
4. Concomitant uncontrolled disease;
5. A diagnosis of bronchiectasis, sarcoidosis, interstitial lung disease, or idiopathic pulmonary fibrosis;
6. Participation in other non-interventional observational trials that might, in the investigator's opinion, influence the assessment for the current study, or participation in any observational or clinical trial in the last 30 days prior to inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients >= 18 y.o. with moderate to severe COPD who are eligible for BREZTRI therapy
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Change in COPD Assessment Test (CAT) score | 24 weeks
  Change from baseline to 24 weeks in the CAT score. Minimum value - "0", maximum value - "5". Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Change in COPD Assessment Test (CAT) score | 12 weeks
  Change from baseline to 12 weeks in the CAT score. Minimum value - "0", maximum value - "5". Higher scores mean worse outcome.
Change in FEV1 | 24 weeks
  Change from baseline to 24 weeks in FEV1
Change in the Treatment Satisfaction Questionnaire for Medication (TSQM) score | 24 weeks
  Change from baseline to 24 weeks in the TSQM score. Minimum score - "1", maximum score - "7". Higher scores mean better outcome.
MCID >= 2 | 24 weeks of treatment
  • Percent of responders using the CAT who achieved MCID (minimal clinically important difference) = 2 or more points after 24 weeks of treatment
>= 20 points at MARS | 24 weeks
  Percent of patients who are high adherent to therapy (who received 20 or more points at MARS) during 24 weeks;
PGI-C - any improvement | 24 weeks of treatment
  Percent of patients with response (any category better than "no change") at the PGI-C after 24 weeks of treatment
PGI-S - change from baseline | after 24 weeks of treatment
  • Percent of patients with change from baseline (before Breztri treatment start) in the severity of general COPD symptoms at the PGI-S after 24 weeks of treatment
To describe treatment safety by AE (adverse events) monitoring | AEs will be collected from the day when the informed consent has been signed (Visit 0) until the time last visit (Visit 2- 24 (+2) weeks after index date) has occurred
  to monitor AE frequency
Treatment safety by AE monitoring | AEs will be collected from the day when the informed consent has been signed (Visit 0) until the time last visit (Visit 2- 24 (+2) weeks after index date) has occurred
  to collect information on treatment discontinuation due to AE

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Research Site, Blagoveshchensk
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Volgograd
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00097&attachmentIdentifier=00ade59f-8ba5-4531-99fa-3a77f455962d&fileName=D5980R00097_Redacted_CSR_Synopsis.pdf&versionIdentifier=